CLINICAL TRIAL: NCT06928532
Title: Seated Tai Chi Improves Dynamic Finger Pointing Task and Sitting Balance Control in Subjects With Parkinson's Disease: A Prospective Study
Brief Title: Seated Tai Chi Improves Dynamic Finger Pointing Task and Sitting Balance Control in Subjects With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.2019/1002
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease and Parkinsonism; Tai Chi
Keywords: Eye-hand coordination; Sitting balance control; Tai Chi; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seated TC (Experimental): Type of intervention: 12-form Yang-style seated Tai Chi routine23 under the supervision and guidance of a certified Tai Chi master Duration: 3 months (24 sessions in total) Frequency: 2 sessions per week, 1 hour per session
  Interventions: Behavioral: Seated TC
- Control (No Intervention): Control group continued with their usual daily routines and activities

INTERVENTIONS:
Behavioral: Seated TC — 3-month seated Tai Chi training (24 sessions in total) given to Parkinson's disease patients
  Arms: Seated TC

SUMMARY:
The goal of this prospective study is to investigate the effects of 3 months seated Tai Chi (TC) practice on the eye-hand coordination and sitting balance control of subjects with Parkinson's disease. The main objective it aims to answer are the effects of seated TC training on:

* Shoulder joint range of motion;
* Eye-hand coordination;
* Dynamic sitting balance control; and
* Quality of life in individuals with Parkinson's disease

Researchers compared seated TC training with a control group to see if it improved the aforementioned outcomes.

Participants completed:

* 3-month TC training of 24 sessions in total
* two sessions per week and each session lasted for 1-hour
* went on with their usual physical activities and routines outside the training

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's disease (PD)
* Mini-Mental State Examination (MMSE) scored over 24
* Individuals with mobility levels suitable for participation in seated TC

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Shoulder mobility | Immediate after 3-month training period
  Shoulder flexion range of motion
Eye-Hand Coordination Test | Immediate after 3-month training period
  Reaction time, movement time, accuracy
Dynamic sitting balance | Immediate after 3-month training period
  Participants were assessed using the Sequential Weight Shifting Test where they were seated on a force platform equipped with four load cells capable of measuring forces ranging from 40 to 400 pounds to calculate their accuracy of centre of pressure shifts during the test
Quality of life of Parkinson's disease patients | Immediate after 3-month training period
  Parkinson's Disease Questionnaire-39 (PDQ-39)

CONTACTS AND LOCATIONS:
Overall Officials: William Wai Nam Tsang, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data is available on reasonable request

DOCUMENTS (1):
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT06928532/ICF_000.pdf